CLINICAL TRIAL: NCT02213406
Title: Fat and the Brain-Neuronal and Sensory Fat Perception
Brief Title: Neuronal and Sensory Perception of Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sabine Frank, Dr., University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: NSFP
Record Dates: First submitted 2014-08-05; First posted 2014-08-11 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Fat Perception in the Brain
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention group (Experimental): Fat detection threshold test, intake of high and low fat yogurt, fMRI-measurements
  Interventions: Dietary Supplement: yogurt

INTERVENTIONS:
Dietary Supplement: yogurt — Subjects will receive yogurt with varying fat concentrations

SUMMARY:
This project will examine neuronal and sensory fat perception. Our hypothesis is that subjects being either hypersensitive or hyposensitive for fat will show different brain activities. Therefore the investigators will conduct functional magnetic resonance imaging (fMRI) and fat detection threshold tests examining neuronal and sensory fat perception.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* lactose intolerance
* fMRI contraindications (metal implants,...)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Fat detection thresholds | each measurement day
  A sensory test will be conducted to establish individual fat detection thresholds. It is expected that subjects* brain activity is dependent on sensory fat sensitivity.

SECONDARY OUTCOMES:
Brain activity | pre and post meal intake
  We are interested in brain activations following the consumption of yogurt with either a high or a low fat concentration. To assess this, before as well as after fat intake brain activity will be measured using functional magnetic resonance imaging (fMRI). We expect that brain activity will differ between the high and the low fat yogurt condition.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, fMEG Center, Tübingen, Germany